CLINICAL TRIAL: NCT05963750
Title: Assessment of the Impact of Virtual Reality on Patient Anxiety During Dental Avulsions Under Local Anesthesia
Acronym: REVIDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-0188
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Tooth Avulsion; Anxiety
Keywords: virtual reality; oral surgery; anxiety
MeSH Terms: conditions — Tooth Avulsion; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A list with numbers from 1 to 120 was produced prior to the study on Excel. Each number was assigned a random group (with and without VR).
  During the first consultation, the patient was assigned a number (the practitioner followed the list on Excel) and therefore a group. Both practitioner and patient knew the patient's group for the next appointment.
  When the patient filled out the questionnaires, he was referring to his assigned number and not his name. Then, the practitioner filled in the Excel file with the data collected (characteristics of the patients, STAI-YA score, VAS), which were associated with the patient's number, and which were therefore anonymous.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality during the surgery (Experimental): Group with the use of virtual reality during the surgery
  Interventions: Other: virtual reality
- control (No Intervention): Group without the use of virtual reality during the surgery

INTERVENTIONS:
Other: virtual reality — virtual reality
  Arms: virtual reality during the surgery

SUMMARY:
Fear of the dentist is a very common phenomenon which delays consultations and brings negative consequences on oral and general health. Virtual reality (VR) reduces children's pain and anxiety during dental care or oral surgery. The aim of this prospective, randomized and controlled study is to show the effectiveness of virtual reality to reduce anxiety in a sample of adults during tooth avulsions under local anesthesia. There is a group with virtual reality and a control group without virtual reality.

Patients complet the State Trait Anxiety Inventory - State - (STAI-YA) questionnaire and the visual analog anxiety scale (VAS) just before and just after the surgery by transcribing the anxiety they feel during it. The main judgement criterion is the evolution of the STAI-YA score before vs during the surgery. Secondary criteria are the relevance of the chosen metric by comparing it to the VAS, defining the factors influencing the evolution of the anxiety score, studying the side effects of VR and the wish to repeat the experience.

DETAILED DESCRIPTION:
The virtual reality experience consisted of putting on a headset with music and a 3D helmet on the eyes that broadcast a landscape in motion (a walk).

The inclusion took place in the University Hospital of Caen between november 2021 and may 2022.

119 patients were randomized into two groups, one with VR and another one without VR. At the end, 105 patients were analyzed.

The main objective was to find a reduction in the STAI-YA score of more than 8 points between before and during the intervention. This analysis was performed in both groups.

During the initial consultation, questions were asked about the medical file and informed consent was sought. Patients were then randomised to one of two groups.

During the second consultation, a STAI-YA questionnaire and a VAS scale were completed, then the intervention was performed with or without virtual reality, depending on the group, and the STAI-YA questionnaire and the VAS scale were again completed by recalling the stress experienced during the surgery.

ELIGIBILITY:
Inclusion Criteria:

- Adults (> 18 years old) coming for at least two dental extractions under local anesthesia

Exclusion Criteria:

* patients suffering of motion sickness,
* claustrophobia,
* uncontrolled epilepsy,
* visual impairment,
* hearing disability,
* non-French speakers,
* pregnant women,
* protected adults
* people followed by a psychiatrist whether for depression, bipolarity, schizophrenia
* The day of the intervention, patients who had consumed anxiolytics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
effectiveness of virtual reality on anxiety (STAI-YA) | Baseline and during the procedure.
  The patient completes two anxiety questionnaires (STAI-YA ) before and during the procedure.
effectiveness of virtual reality on anxiety (Visual Analogue Scale) | Baseline and during the procedure.
  The patient completes two anxiety questionnaires (Visual Analogue Scale) before and during the procedure.

SECONDARY OUTCOMES:
Comparability of the results with another metric for assessing anxiety | 1 day of surgery
  The difference in the visual analogue anxiety scale score between before and during surgery was studied. A reduction of 2cm was sought.
factors influencing changes in the STAI-YA anxiety score | 1 day of surgery
  Using the completed medical records (age, sex, smoking habits, etc.) we looked for any factors influencing the results.
The wish to renew the virtual reality experience | 1 day of surgery
  the question "would you like to repeat the experience for other dental avulsions" was asked to the group who had benefited from virtual reality

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Veyssiere, M.D, Study Director — CHU CAEN
Locations (1):
- CHU Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No
this is not planned